CLINICAL TRIAL: NCT00001056
Title: A Phase I Multicenter Clinical Trial to Evaluate the Safety and Immunogenicity of Vaccinia Derived HIV-1 Recombinant Envelope Glycoprotein (gp160) of Human Immunodeficiency Virus: Evaluation of a 200-mcg Dose
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immuno-US (Industry)
Responsible Party: Sponsor
Masking: Double | Purpose: Prevention
Other Study IDs: AVEG 004A; 10544 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; Vaccinia Virus; Viral Vaccines; HIV-1; HIV Envelope Protein gp160; AIDS Vaccines; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections; Vaccinia

INTERVENTIONS:
Biological: gp160 Vaccine (Immuno-AG)

SUMMARY:
To determine the safety of and immune response to vaccinia-derived HIV-1 recombinant envelope glycoprotein (gp160) at a dose of 200 mcg in human volunteers; to evaluate duration of antibody response and its relationship to the dose and frequency of inoculation.

Although recent advances have been made in antiviral therapy against AIDS, there is currently no cure for AIDS. It is likely that the ultimate control of the disease depends on the development of safe and effective vaccines against HIV.

DETAILED DESCRIPTION:
Although recent advances have been made in antiviral therapy against AIDS, there is currently no cure for AIDS. It is likely that the ultimate control of the disease depends on the development of safe and effective vaccines against HIV.

Healthy, adult volunteers without identifiable high-risk behavior for HIV-1 infection are randomly assigned to receive three injections of either 200 mcg gp160 vaccine or a placebo. At each participating site, four volunteers receive vaccine and two volunteers receive placebo. Primary immunization and two booster immunizations at day 30 and day 180 are done in an outpatient setting. Volunteers are closely monitored for the first 2 weeks postimmunization (primary and boosters), and extensively followed for 2 years. Volunteers may be offered an additional booster of the same preparation at 12 months.

ELIGIBILITY:
Inclusion Criteria

Patients must be:

* Normal, healthy, HIV-negative adults who fully comprehend the purpose and details of the study.
* Available for 2 years of follow-up.

Exclusion Criteria

Co-existing Condition:

Patients with the following conditions or symptoms are excluded:

* History of positive PPD (tuberculin test) and abnormal chest x-ray.
* Positive syphilis serology (e.g., RPR).
* Positive for circulating hepatitis B surface antigen.

Patients with the following are excluded:

* They or their sexual partners have identifiable high-risk behavior for HIV infection.
* History of immunodeficiency or chronic illness.
* Evidence of psychological or psychiatric problems that may lead to noncompliance.

Prior Medication:

Excluded:

* Immunosuppressive medications.

Prior Treatment:

Excluded:

* Blood transfusions or cryoprecipitates within the past 6 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Study Completion 1994-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Belshe R, Study Chair
Locations (3):
- United States (3):
  - St. Louis Univ. School of Medicine AVEG, St Louis, Missouri
  - Univ. of Rochester AVEG, Rochester, New York
  - Vanderbilt Univ. Hosp. AVEG, Nashville, Tennessee

REFERENCES:
- [Background] Keefer MC, Wolff M, Gorse GJ, Graham BS, Corey L, Clements-Mann ML, Verani-Ketter N, Erb S, Smith CM, Belshe RB, Wagner LJ, McElrath MJ, Schwartz DH, Fast P. Safety profile of phase I and II preventive HIV type 1 envelope vaccination: experience of the NIAID AIDS Vaccine Evaluation Group. AIDS Res Hum Retroviruses. 1997 Sep 20;13(14):1163-77. doi: 10.1089/aid.1997.13.1163. PMID 9310283